CLINICAL TRIAL: NCT03164083
Title: Evaluation the Effects of Intra-articular Injection of Mesenchymal Stem Cells and Stromal Vascular Fraction Patients With Knee Joint Osteoarthritis, Triple Blind Randomized Clinical Trial
Brief Title: The Effects of Stromal Vascular Fraction and Mesenchymal Stem Cells as Intra-articular Injection in Knee Joint Osteoarthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: not approved by sponsor
Sponsor: SCARM Institute, Tabriz, Iran (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SCARM-Osteoarthritis-001
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2019-01

CONDITIONS: Osteoarthritis
Keywords: Joint Diseases; Musculoskeletal Diseases; Arthritis
MeSH Terms: conditions — Osteoarthritis; Joint Diseases; Musculoskeletal Diseases; Arthritis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mesenchymal stem cell (Experimental): Patients with knee joint osteoarthritis who underwent intra articular mesenchymal stem cell injection
  Interventions: Biological: Mesenchymal stem cell
- placebo (Experimental): The patients who are in control group and underwent placebo injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Mesenchymal stem cell — intra articular injection of mesenchymal stem cell Other Name: stem cell transplantation
  Arms: mesenchymal stem cell
Biological: Placebo — Patients with knee joint osteoarthritis who underwent intra articular placebo injection
  Arms: placebo

SUMMARY:
Osteoarthritis of the knee is one of the most common causes of disability among elderly. As the disease progresses the cartilage become frustrated, surrounding bone react to become thicker and inflammation occurs in subchondral bone seen in T2-weighted MRI as increase in signal density. Patients are treated initially by pain management. In patients who don't response to first line treatment invasive treatment like total knee replacement is done. The investigators designed this clinical study with the aim of evaluating therapeutic effects of intra-articular injection of bone marrow Mesenchymal Stem Cells (MSC) and stromal Vascular Fraction (SVF) in patients with severe knee osteoarthritis

DETAILED DESCRIPTION:
This is single center, randomized, triple blind phase II clinical study. Patients will be divided into two groups of case and control. All subjects will undergo bone marrow aspiration. Mesenchymal Stem Cells will be isolated from bone marrow and stromal Vascular Fraction fram lipoaspirate, cultured and transplanted back to the knee joint. Patients of case group will receive cell injection 1 and 4 months after bone marrow aspiration. Placebo will be administered in this group 6 months after the first injection. Patients of control group will receive placebo 1 and 4 months after bone marrow aspiration. They all receive cell injection 6 months after first placebo injection. Follow up visit will occur at 2 and 6 weeks, and 3 and 6 months after the first injection. Radiological exams will be performed before and 6 months after the first injection by MRI. Clinical quantitative assessment will measure joint function by the WOMAC index and pain by the visual analogue scale

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis diagnosed by MRI

Exclusion Criteria:

* Pregnancy or lactating
* Positive tests for HIV, Hepatitis C virus (HCV), Hepatitis C virus (HBV)
* Active neurologic disorder
* End organ damage
* Uncontrolled endocrine disorder

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-10 (Estimated); Primary Completion 2020-08-21 (Estimated); Study Completion 2020-12-05 (Estimated)

PRIMARY OUTCOMES:
physical function improvement | 2 weeks
  Evaluation the physical function improvement Measured by WOMAC osteoarthritis index after cell injection
Change in pain density | 2 weeks
  Evaluation the changing of pain density measured by Visual Analogue Scale after cell injection

SECONDARY OUTCOMES:
Joint swelling | 3 months
  Evaluation the joint swelling by physical examination after intra articular cell injection
Joint erythema | 3 months
  Evaluation the joint erythema by physical examination after cell injection
Deterioration of joint function | 3 months
  Evaluation the deterioration of joint function by physical examination after intra articular cell injection
Allergic reactions | 3 months
  Evaluation the allergic reactions like skin rash,skin erythema, dyspnea by physical examination after cell injection

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nouri, Ph.D, Study Chair — Head of SCARM Institute; Peyman Keyhanvar, MD, Ph.D, Study Director — Deputy for translational medicine of SCARM institute; Seyed Kazem Shakouri, Physiatrist, Principal Investigator — Tabriz University of Medical Sciences; Neda keyhanvar, Ph.D, Principal Investigator — SCARM institute; Sepideh Bastani, MSc, Principal Investigator — SCARM institute
Locations (1):
- SCARM Institute, Tabriz, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pak J, Lee JH, Park KS, Park M, Kang LW, Lee SH. Current use of autologous adipose tissue-derived stromal vascular fraction cells for orthopedic applications. J Biomed Sci. 2017 Jan 31;24(1):9. doi: 10.1186/s12929-017-0318-z. PMID 28143470
- [Result] Pak J, Lee JH, Kartolo WA, Lee SH. Cartilage Regeneration in Human with Adipose Tissue-Derived Stem Cells: Current Status in Clinical Implications. Biomed Res Int. 2016;2016:4702674. doi: 10.1155/2016/4702674. Epub 2016 Jan 6. PMID 26881220
- [Result] Koh YG, Choi YJ, Kwon SK, Kim YS, Yeo JE. Clinical results and second-look arthroscopic findings after treatment with adipose-derived stem cells for knee osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2015 May;23(5):1308-1316. doi: 10.1007/s00167-013-2807-2. Epub 2013 Dec 11. PMID 24326779
- [Result] Pires de Carvalho P, Hamel KM, Duarte R, King AG, Haque M, Dietrich MA, Wu X, Shah F, Burk D, Reis RL, Rood J, Zhang P, Lopez M, Gimble JM, Dasa V. Comparison of infrapatellar and subcutaneous adipose tissue stromal vascular fraction and stromal/stem cells in osteoarthritic subjects. J Tissue Eng Regen Med. 2014 Oct;8(10):757-62. doi: 10.1002/term.1565. Epub 2012 Jul 16. PMID 22807102